CLINICAL TRIAL: NCT02601456
Title: The Effect of Prolonged Effort on the Bilateral Asymmetry in Trans Tibial Amputee Running With Running Specific Prosthesis
Brief Title: Changes in Trans Tibial Amputee Running Asymmetry During Prolonged Effort
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-14-1834-ISN-CTIL
Record Dates: First submitted 2015-11-05; First posted 2015-11-10 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-01

CONDITIONS: Amputation, Traumatic
Keywords: Amputation, Traumatic; Biomechanics; Asymmetry; Amputee Running; Prolonged Effort
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the effect of prolonged effort in long distance running on the biomechanical bilateral asymmetry in the lower limbs of trans tibial amputee running with running specific prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral traumatic trans tibial amputee.
* Experience in running with running specific prosthesis.
* Ability to run for at least 20 minutes.

Exclusion Criteria:

* Injury or other orthopedic or neurologic issue that compromises the gait.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The changes in step length asymmetry after prolonged effort in running on a treadmill. | Several measurements during 20-30 minutes run.
  Step length will be recorded by the v-gait analysis system during the running test for 20 seconds at certain points of the run: minute 0, 5, 10, 15, 20, 25, 30. If the subject will ask to stop the run, 20 seconds will be recorded prior to the termination of the run.
The changes in contact time asymmetry after prolonged effort in running on a treadmill. | Several measurements during 30 minutes run.
  Contact time will be recorded by the v-gait analysis system during the running test for 20 seconds at certain points of the run: minute 0, 5, 10, 15, 20, 25, 30. If the subject will ask to stop the run, 20 seconds will be recorded prior to the termination of the run.
The changes in flight time asymmetry after prolonged effort in running on a treadmill. | Several measurements during 30 minutes run.
  Flight time will be recorded by the v-gait analysis system during the running test for 20 seconds at certain points of the run: minute 0, 5, 10, 15, 20, 25, 30. If the subject will ask to stop the run, 20 seconds will be recorded prior to the termination of the run.
The changes in hip angles asymmetry after prolonged effort in running on a treadmill. | Several measurements during 30 minutes run.
  Hip angles will be recorded by the v-gait analysis system during the running test for 20 seconds at certain points of the run: minute 0, 5, 10, 15, 20, 25, 30. If the subject will ask to stop the run, 20 seconds will be recorded prior to the termination of the run.
The changes in knee angles asymmetry after prolonged effort in running on a treadmill. | Several measurements during 30 minutes run.
  Knee angles will be recorded by the v-gait analysis system during the running test for 20 seconds at certain points of the run: minute 0, 5, 10, 15, 20, 25, 30. If the subject will ask to stop the run, 20 seconds will be recorded prior to the termination of the run.
The changes in vertical ground reaction force asymmetry after prolonged effort in running. on a treadmill | Several measurements during 30 minutes run.
  Vertical ground reaction force will be recorded by the v-gait analysis system during the running test for 20 seconds at certain points of the run: minute 0, 5, 10, 15, 20, 25, 30. If the subject will ask to stop the run, 20 seconds will be recorded prior to the termination of the run.
The changes in ground reaction impulse asymmetry after prolonged effort in running on a treadmill. | Several measurements during 30 minutes run.
  Vertical ground reaction impulse will be recorded by the v-gait analysis system during the running test for 20 seconds at certain points of the run: minute 0, 5, 10, 15, 20, 25, 30. If the subject will ask to stop the run, 20 seconds will be recorded prior to the termination of the run.

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Ziev-Ner, Dr., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel